CLINICAL TRIAL: NCT04398992
Title: Chinese Registry of Additive Anti-inflammatory Action for Aortopathy & Arteriopathy (5A) Protocol: Rationale, Design and Methodology
Brief Title: Additive Anti-inflammatory Action for Aortopathy & Arteriopathy
Status: Recruiting | Type: Observational
Sponsor: Nanjing Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Hong Liu, Investigator of Department of Cardiac Surgery, Nanjing Medical University
Other Study IDs: 5A-Plan
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Aortic Syndrome
Keywords: Acute Aortic Syndrome
MeSH Terms: conditions — Acute Aortic Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — Data were collected by a designed form. Statistic software was used to analyze clinical data.

SUMMARY:
Acute aortic syndrome (AAS) is a life-threatening condition. Inflammation plays a key role in the pathogenesis, development and progression of AAS, and is associated with significant mortality and morbidity. Understanding the inflammatory responses and inflammation resolutions is essential for an appropriate management of AAS.

Twenty Chinese cardiovascular centers have collaborated to create a multicenter observational registry (named Chinese registry of Additive Anti-inflammatory Action for Aortopathy & Arteriopathy [5A]), with consecutive enrollment of adult patients who underwent surgery for AAS that was started on Jan 1, 2016 and will be ended on December 31, 2040. Specially, the impact of inflammation and anti-inflammatory strategies on the early and late adverse events are investigated. Primary outcomes are severe systemic inflammatory response syndrome (SIRS), multiple organ dysfunction syndrome (MODS), Sequential Organ Failure Assessment (SOFA) scores at 7 days following this current surgery. Secondary outcomes are SISR, 30-day mortality, operative mortality, hospital mortality, new-onset stroke, acute kidney injury, surgical site infection, reoperation for bleeding, blood transfusion and length of stay in the intensive care unit.

DETAILED DESCRIPTION:
Aortopathy represent a major clinical challenge and are regarded as one of the leading causes of mortality among cardiovascular disorders. However, the pathological mechanisms underlying aortopathy are still far from being well understood, which makes treating this life-threatening challenging. It is increasingly clear that inflammation plays a key role in the development and progression of acute aortic syndrome (AAS) independent of cholesterol and other traditional risk factors, and characterizes both systemic and local condition.

Currently, surgery is considered the best treatment option for patients with AAS. In addition to systemic inflammatory responses triggered by AAS itself, however, procedural factors including surgical trauma, anesthesia, cardiopulmonary bypass, hypothermia, circulatory arrest, and blood transfusion as well as mechanical ventilation initiated a cascade of inflammation, which further exacerbates "inflammatory storm", and is associated with significant postoperative mortality and morbidity. Along with surgical evolutions, scientists have made new discoveries and achievements in the underlying mechanism and understanding of inflammation of AAS, which greatly encourage us to optimize treatment for these patients. Going beyond traditional surgery, anti-inflammatory action is crucially important to target the residual cardiovascular risk by specific anti-inflammatory interventions as a crucially adjunct therapeutic strategy to improve the well-being of patient.

A better understanding of the interaction between patient's inflammatory responses and anti-inflammatory strategies which may limit the residual cardiovascular risk is essential for the development of novel preventive, diagnostic, and therapeutic approaches, providing a critical pathophysiological insight into the role of inflammation in risk assessment and anti-inflammatory targeting. The epidemiological observation that biomarkers of inflammation are associated with clinical cardiovascular risk supports the theory that targeted anti-inflammatory treatment appears to be a promising strategy in reducing residual cardiovascular risk on the background of traditional surgical repair as well as basic therapy. Previous researches have shown that ulinastatin used in cardiac surgery may be effective in prevention of cardiovascular events through an anti-inflammatory effect. This residual inflammatory risk has increasingly become a viable therapeutic targeting on the background of validated surgical repair as well as basic medical therapy for AAS.

Although aortic dissection registries have been established during the last years, such as the International Registry of Acute Aortic Dissection (IRAD), the Nordic Consortium for Acute Type A Aortic Dissection (NORCAAD) Registry, German Registry for Acute Aortic Dissection type A (GERAADA), the Society of Thoracic Surgeon (STS) database , and European Registry of Type A Aortic Dissection (ERTAAD), there are currently no dedicated registry to prospective collections and characteristics of inflammatory responses, anti-inflammatory strategies, and clinical outcomes especially for AAS patients. We have established a multicenter research collaboration (named "Chinese Registry of Additive Anti-inflammatory Action for Aortopathy & Arteriopathy [5A]") and planned a prospectively observational study to understand the patient's inflammatory responses, characterize the potential anti-inflammatory strategies, and evaluate clinical outcome and prognosis of AAS patients at 15 years in a large study of Chinese population.

ELIGIBILITY:
Inclusion criteria

* Aged 18 years or older.
* Patients with diagnosis of AAS, including aortic dissection, penetrating aortic ulcer or intramural hematoma.
* Symptoms started within 14 days from surgery.
* Patients received medical therapy, open surgical, endovascular, or hybrid repair.
* Any other major cardiac surgical procedure concomitant with surgery for AAS, such as coronary artery bypass grafting or carotid artery replacement;
* The patient or guardian agrees to participate in this study. Exclusion criteria
* Patients aged < 18 years.
* Onset of symptoms > 14 days from surgery.
* AAS secondary to traumatic or iatrogenic injury.
* Patients who declined participation in registration and follow-up investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients suffering AAS
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Operative mortality | 30 days after treatment
  Operative mortality was defined as any death, regardless of cause, occurring whether within 30 days after surgery in or out of the hospital or after 30 days during the same hospitalization subsequent to the operation.
Severe systemic inflammatory response syndrome (SIRS) | 7 days after treatment
  SIRS was defined as the presence of at least 2 of the 4 age-specific criteria: temperature, heart rate, respiratory rate, and leukocyte count, one of which must be abnormal temperature or leukocyte count. severe SIRS was defined as meeting all 4 aforementioned criteria, measured immediately following surgery through postoperative day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Hong-jia Zhang, MD, Study Director — Beijing Anzhen Hospital; Hong Liu, Principal Investigator — Nanjing Medical University; Si-chong Qian, Principal Investigator — Beijing Anzhen Hospital
Locations (34):
- China (34):
  - Beijing Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing Hospital of Jiangsu Provincial People's Hospital, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - QianXiNan People's Hospital, Xingyi, Guizhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Third Affiliated Hospital of Soochow University, Changzhou, Jiangsu
  - Suqian Hospital of of Nanjing Medical University, Suqian, Jiangsu
  - Dongtai People's Hospital, Yancheng, Jiangsu
  - Subei People's Hospital of Jiangsu Province, Yangzhou, Jiangsu
  - the Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai DeltaHealth Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Seventh Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Friendship Hospital of Yili Kazak Autonomous Prefecture, Yining, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Anzhen Hospital Capital Medical University, Beijing
  - Beijing Chaoyang Hospital, Beijing
  - the First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Xiangya Hospital Central South University, Changsha
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - the First Affiliated Hospital of Guilin Medical College, Guilin
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Nanjing First Hospital, Nanjing Medical University, Nanjing
  - the Affiliated Hospital of Qingdao University, Qingdao
  - Shanghai East Hospital Tongji University, Shanghai
  - the First Affiliated Hospital of Shantou University Medical College, Shantou
  - Teda International Cardiovascular Hospital, Tianjin
  - Tianjin Chest Hospital, Tianjin
  - Xiamen Cardiovascular Hospital, Xiamen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu H, Li HY, Li YL, Wu Y, Gu JX, Diao YF, Shao YF, Sun LZ, Qian SC, Zhang HJ; 5A Investigators. Operative Mortality After Type A Aortic Dissection Surgery: Differences Based on Sex and Age. JACC Adv. 2024 Mar 14;3(4):100909. doi: 10.1016/j.jacadv.2024.100909. eCollection 2024 Apr. PMID 38939657
- [Derived] Liu H, Diao YF, Shao YF, Qian SC, Zeng ZH, Fan GL, Ma LY, Zhang HJ; on the behalf of the Additive Anti-inflammatory Action for Aortopathy & Arteriopathy (5A) Investigators. Prognostic implication of residual inflammatory trajectories in acute type I aortic dissection: dual-center prospective cohort study. Int J Surg. 2024 Jun 1;110(6):3346-3356. doi: 10.1097/JS9.0000000000001245. PMID 38445499
- [Derived] Liu H, Qian SC, Li HY, Shao YF, Zhang HJ; China Additive Anti-inflammatory Action for Aortopathy, Arteriopathy (5A) Investigators. Chinese Additive Anti-inflammatory Action for Aortopathy & Arteriopathy (5A) Registry protocol: rationale, design and methodology. BMC Cardiovasc Disord. 2024 Feb 21;24(1):120. doi: 10.1186/s12872-024-03760-y. PMID 38383323
- [Derived] Liu H, Sun BQ, Qian SC, Sun MY, Shao YF, Ding Y, Li H, Zhang HJ. Contemporary use and outcome of Cabrol shunt in type A aortic dissection surgery: insight from China 5A study. Open Heart. 2023 Dec 9;10(2):e002465. doi: 10.1136/openhrt-2023-002465. PMID 38070883
- [Derived] Zhao HL, Tang ZW, Diao YF, Xu XF, Qian SC, Li HY, Shao YF, Zhao S, Liu H; on the behalf of the Additive Anti-inflammatory Action for Aortopathy, Arteriopathy (5A) Investigators. Inflammatory profiles define phenotypes with clinical relevance in acute type A aortic dissection. J Cardiovasc Transl Res. 2023 Dec;16(6):1383-1391. doi: 10.1007/s12265-023-10436-z. Epub 2023 Sep 15. PMID 37713048